CLINICAL TRIAL: NCT01016353
Title: A Prospective Study Examining Clinical Outcomes Associated With the Management of the Open Abdomen With the ABThera™ Open Abdomen Negative Pressure Therapy System and Barker's Vacuum Packing Technique
Brief Title: Open Abdomen Study Comparing ABThera™ Open Abdomen Negative Pressure Therapy System and Barker's Vacuum Packing Technique
Status: Completed | Type: Observational
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Other Study IDs: ABT2009-50
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Open Abdomen
Keywords: ABThera; Barker's Vacuum Packing Technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: NPWT — ABThera Open Abdomen Negative Pressure Therapy System
  Other Names: ABThera
Device: BVPT — Barker's Vacuum Packing Technique

SUMMARY:
This study is being done to gather data that will be used to compare two different TAC (Temporary Abdominal Closure) methods that your doctor may use. The two TAC methods being compared are the Barker's vacuum packing technique or BVPT and the Open Abdomen Negative Pressure Therapy System (ABThera) developed by the sponsor of this research (KCI, San Antonio, TX). The BVPT is made up of supplies that are stocked in most surgery rooms. The ABThera dressing is available commercially. Neither method will be supplied to the doctor (Principal Investigator), so that in no way would the subject's standard of care be different from what they would get if the study was not being done.

This study is observational and only collects data about how the subject progresses after surgery TAC is used. When a study is observational it means that the subject's standard medical care will not be altered in any way, simply watched. The doctor will not change treatment of your open abdomen.

DETAILED DESCRIPTION:
This study is being done to gather data that will be used to compare two different TAC (Temporary Abdominal Closure) methods. The two TAC methods being compared are the Barker's vacuum packing technique or BVPT and the Open Abdomen Negative Pressure Therapy System (ABThera) developed by the sponsor of this research (KCI, San Antonio, TX). The BVPT is made up of supplies that are stocked in most surgery rooms. The ABThera dressing is available commercially. Neither method will be supplied to the doctor (Principal Investigator), so that in no way would the subject's standard of care be different from what they would get if the study was not being done.

This study is observational and only collects data about how the subject progresses after surgery TAC is used. When a study is observational it means that the subject's standard medical care will not be altered in any way, simply watched. The doctor will not change treatment of your open abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18-75 years of age
2. OA Subjects treated with only one of the following TACs at initial placement (defined as the time of the first application of a TAC method):

   1. ABThera
   2. BVPT

Exclusion Criteria:

1. Pregnant females
2. Active, uncontrolled hemorrhage at the time of TAC placement
3. Diagnosis of pre-existing bleeding disorder
4. Known allergy or hypersensitivity to polyvinyl, polyurethane, acrylic, or acrylic adhesive
5. Subjects with fistulas
6. Subjects who have been enrolled in this study previously
7. Documented history of Child-Pugh Turcot Liver Dysfunction - Class C (10-15 points) at the time of enrollment
8. Subjects with body mass index (BMI) > 40 as estimated at the time of Emergency Department (ED) or OR admission
9. Known New York Heart Association Functional Classification - Class IV at the time of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergent Care
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of South Alabama Medical Center, Mobile, Alabama
  - LAC/USC Medical Center, Los Angeles, California
  - Orlando Regional Medical Center, Orlando, Florida
  - Cook County Medical Center, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryand, Baltimore, Maryland
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Regional Medical Center, Memphis, Tennessee

REFERENCES:
- [Derived] Bjorck M, Kirkpatrick AW, Cheatham M, Kaplan M, Leppaniemi A, De Waele JJ. Amended Classification of the Open Abdomen. Scand J Surg. 2016 Mar;105(1):5-10. doi: 10.1177/1457496916631853. Epub 2016 Feb 29. PMID 26929286

RESULTS

PARTICIPANT FLOW:
Groups:
- BVPT: Barker's vacuum-packing technique (BVPT)
Period: Overall Study
Arm/Group | NPWT | BVPT
Started | 180 | 103
Completed | 178 | 102
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPWT | BVPT | Total
Number analyzed (Participants) | 178 | 102 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (17) | 39 (16) | 40 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 142 | 74 | 216
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian | 1 | 1 | 2
  Race/Ethnicity: Asian | 4 | 3 | 7
  Race/Ethnicity: Black or African American | 54 | 40 | 94
  Race/Ethnicity: Hispanic or Latino | 37 | 10 | 47
  Race/Ethnicity: Native Hawaiian | 1 | 1 | 2
  Race/Ethnicity: White | 81 | 47 | 128
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 178 | 102 | 280

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Fascial Closure
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | NPWT | BVPT
Number analyzed (Participants) | 178 | 102
Participants | 139 | 69
Statistical Analysis 1: Comparison: NPWT vs BVPT; Test type: Superiority; p = 0.06, Log Rank

ADVERSE EVENTS:
Time Frame: 30 day
Description: All-cause mortality was an endpoint for the study, therefore it was reported based on the mITT population rather than the safety population. mITT population included subjects who received any study-related TAC, regardless of its duration, had a valid baseline, and at least 1 post baseline assessment for any of the study efficacy parameters.
Arm/Group | NPWT | BVPT
All-Cause Mortality (participants affected / at risk) | 21/178 | 20/102
Serious Adverse Events (participants affected / at risk) | 3/180 | 0/103
Other Adverse Events (participants affected / at risk) | 65/180 | 36/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NPWT (N=180) | BVPT (N=103)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NPWT (N=180) | BVPT (N=103)
Abdominal Adhesions (Gastrointestinal disorders) | 9 | 6
Abdominal Infection (Infections and infestations) | 10 | 10
Gastrointestinal Necrosis (Gastrointestinal disorders) | 12 | 2
Intra-Abdominal Hypertension (Gastrointestinal disorders) | 22 | 9
Intraloop Adhesions (Gastrointestinal disorders) | 15 | 1
Loss of Fascial Domain (Musculoskeletal and connective tissue disorders) | 14 | 9
Mulitple Organ Dysfunction Syndrome (General disorders) | 12 | 12
Sepsis (Infections and infestations) | 16 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days